Medication Development for Protracted Abstinence in Alcoholism: Suvorexant Versus Placebo

NCT04229095

Informed Consent Form-02/24/2022



#### SCRIPPS IRB

#### CONSENT TO PARTICIPATE IN RESEARCH

#### Suvorexant for Protracted Abstinence in Alcoholism

PRINCIPAL INVESTIGATOR: Barbara J. Mason, Ph.D.

Professor, Department of Molecular Medicine

Laboratory of Clinical Psychopharmacology, Scripps Research

SUB-INVESTIGATORS:

Jessica Bess, M.S.W. SusanQuello, B.S., B.A. Farhad Shadan, M.D., Ph.D.

Alan Beneze, M.D. Adnan Begovic, M.D.

STUDY CONTACT PERSON: Jessica Bess, M.S.W. (858) 784-7567

**RESEARCH SITE:** 

Scripps Research

Laboratory of Clinical Psychopharmacology

3366 Torrey Pines Court, Suite 305, La Jolla, CA 92037

Before you start reading about this research, please read the California Experimental Subjects' Bill of Rights, which is page 10 of this form.

#### What should I know about this research?

You are being asked to be in a research study to test the effectiveness of suvorexant (Belsomra®) for reducing alcohol cravings. This study requires one overnight stay at the Center for Clinical Research (CCR) located at the Altman Clinical and Translational Research Institute (ACTRI) on the University of California San Diego Health's La Jolla campus. You must not drink alcohol for at least 2 days prior to the overnight stay. To comply with UCSD-ACTRI's "COVID-Free" requirement for overnight visits, you must have a COVID-19 nasal swab test completed 3 days prior to your overnight stay. The study doctor will provide you with a prescription for the test, and it will be your responsibility to complete the test at one of UCSD's drive-thru testing sites for COVID-193 days prior to your second visit. A list of UCSDCOVID-19 testing sites will be provided to you at your first study visit. Your participation in this study is completely voluntary. It is your choice if you want to be in this study. This form will help you decide.

If you agree to join, you can leave the study at any time. If you do not agree to join, or if you leave, you will not be penalized or lose any benefits that you had before starting the study. Take as much time as you need to make your choice and ask the study doctor or staff any questions. If you agree to join, please sign this form after you understand all of the information and your questions have been answered.

Version 02/11/2022 



### Why is this research being done?

This research is being done to find out if suvorexant will help reduce the urge to drink in people with alcohol use disorder. Suvorexant may be a possible treatment to prevent relapse following withdrawal from alcohol.

You have been asked to participate because you may meet criteria for alcohol use disorder and are not currently seeking treatment. Investigators at Scripps Research hope to learn how well suvorexant (a medication used to treat insomnia) works in comparison to a placebo pill for reducing craving for alcohol. This study involves two laboratory sessions at Scripps Research. During the first mini cue laboratory session at the screening visit, you will be asked how much you want to drink. During the second alcohol cue laboratory session you will be asked how much you want to drink while your body responses are being recorded. The second laboratory session will be scheduled between 12:30 p.m. – 3:30 p.m. the day after you have taken a drug that may change your response to alcohol. The drugs to be used in this study are suvorexant or placebo. A "placebo" looks like study drug but does not contain real drug.

Suvorexant is a drug that has not been approved by the US Food and Drug Administration (FDA) to treat alcohol use disorder (but is approved for a different purpose, treatment of insomnia). This study involves a single-dose administration of suvorexant 20 mg or placebo between 12:30 a.m. – 3:30 a.m. during a one-night, inpatient stay at the CCR located at the ACTRI on UC San Diego Health's La Jolla campus. The investigators hope that suvorexant will reduce craving for alcohol in people with alcohol use disorder by helping to normalize their brain activity in early abstinence, thereby reducing craving.

Up to 50people will be admitted to the study, all of them here at Scripps Research and the Center for Clinical Research. To date, 3subjects have been enrolled in this study.

### How long is the study?

If the study suits you and you agree to join, you will be in it over a period of about 2weeks.

### What will happen to me?

You will first come to Scripps Research for a screening visit. During that visit, which will last about 2 hours, you will be asked questions regarding your alcohol use and health. Blood and urine samples will be collected.

At the next visit, a doctor will examine you at Scripps Research. This examination and the medical care you will receive in the study is not the same as seeing your regular doctor. You will also fill out some questionnaires.

Some procedures and tests would be done to determine your eligibility, even if you did not join the study. They are:

- Your medical history
- Your history of alcohol use
- Electrocardiogram (ECG) to measure your heart rate and rhythm
- Urine sample for kidney function, drug screen and pregnancy test (if female)
- Blood sample



These procedures and tests will be repeated at some visits (see visit schedule below):

Blood sample: You will be asked to have a blood sample drawn three times during this study. The medical assistant will draw a blood sample (2-4 teaspoons) from your vein for lab tests of your body functions, and factors related to your alcohol use disorder or response to study procedures, such as the amount of study drug in your blood. Blood samples will be taken at the screening visit (Visit 1), at Visit 2 prior to your overnight stay at the inpatient clinical research unit, and the following afternoon prior to the alcohol cue laboratory session. If you are female, you will also be tested to be sure that you are not pregnant.

Urine sample: You will be asked to give aurine sample to screen for drugs of abuse (Visits 1 and 2) and to verify abstinence from alcohol on Visit 2. If your urine shows you have used any disallowed drugs or alcohol you will not be able to proceed with the study and you will not be paid for the visit. If you are female, you will also be asked to provide a urine sample at Visit 2 for a pregnancy test.

Vital Signs: Your blood pressure, heart rate, temperature and weight (vital signs) will be measured.

**Breath Samples:** Samples of your breath will be collected at each study visit. You will be asked to blow into two small tubes for up to 15 seconds. This is done to measure alcohol and carbon monoxide levels in your body.

ECG: Self-stick pads will be placed on your chest, arms and legs. Wires will be attached to the pads and to a machine that will record the electrical activity of your heart. An electrocardiogram (ECG) is a tracing of your heart's activity. The ECG will be performed at Visit 2.

Medication/Study Drug: If you join the study you will be assigned, by chance, to receive either suvorexant or placebo. You have a 1-in-2 chance of getting real drug. You won't know which you get, and neither will the study physician or staff. The study doctor could find out in an emergency. Study drug will be dispensed at the Center for Clinical Research between 12:30 a.m. – 3:30 a.m. during your overnight visit.

Laboratory Session: During thesecond laboratory session which will occur between 12:30 p.m. – 3:30 p.m. at Scripps Research on the day of inpatient discharge, you will be asked to rate your craving for alcohol following exposure to pictures that may cause different emotions and after viewing and smelling a glass of water and/or your preferred alcoholic beverage (that you are not to drink). In addition to craving, we will also be measuring your heart rate; facial movements and skin responses during that time. You must not drink alcohol for at least 2 days before your medical clearance at Visit #2. A urine sample will be collected to measure ethyl glucuronide and ethyl sulfate (EtG/EtS), which can reliably detect alcohol metabolites in urine for up to 80 hours after drinking alcohol. You will be asked to blow into a small tube for up to 15 seconds to measure breath alcohol on the day of the visit.

Follow Up: A virtual follow-up visit (Visit 3) will be scheduled week after your alcohol laboratory session to make sure you are as healthy as you were at the start of the study. The researcher will tell you about treatment options and offer referral choices if you want treatment.



IRB NUMBER: IRB-19-7450 Scripps IRB APPROVAL DATE: 02/24/2022 IRB EXPIRATION DATE: 02/10/2023

#### Visit Schedule

| Scheduled Procedures Visit | Screeni<br>ng | 2<br>Randomizati<br>on/<br>Overnight<br>stay | Follow-<br>up |
|---|---|---|---|
| Informed consent; demographics; medical and alcohol history; Illicit Drug Use Index; MINI; Alcohol Use Disorder Criteria Fagerstrom Test for Nicotine Dependence | Х | | |
| BAC, vital signs, concomitant treatments | X | X | X. |
| Pregnancy test <sup>1</sup> | X | X | |
| Blood draw for plasma cortisol and drug plasma concentration <sup>2</sup> | | X | |
| Nasal swab test for COVID-193 | | | |
| ECG | | X | |
| Urinalysis, CBC w/diff, blood chemistry | X | | |
| Urine Drug Screen (UDS) | X | X | |
| Urine EtG/EtS | | X | |
| Mini cue session- in vivo beverage presentation | X | | |
| Alcohol cue session | | X | |
| Timeline Follow Back Interview- TLFB Alcohol Craving Questionnaire- ACQ Pittsburg Sleep Quality Index-PSQI Beck Depression Inventory-BDI-II State-Trait Anxiety Inventory-STAI Brief Irritability Test (BITe) | х | Х | Х |
| Physical Exam | | X | X |
| Adverse Events (AE's), Concurrent Drug Therapy | X | X | X |
| Dispense study medication | | X | |
| Overnight, inpatient stay | | X | |
| CIWA | | X | |
| The Epworth Sleepiness Scale | | X | |
| Addiction Research Center Inventory-ARCI Post-Drug Questionnaire | | X | |
| Motivational Interviewing | | | X |

<sup>1 -</sup> Females only. Blood sample at Visit 1 and urine sample at Visit 2.

## Could I experience any side effects or discomforts?

All drugs can cause reactions or side effects. The most common adverse reaction (reported in 5% or more of patients treated with suvorexant and at least twice the placebo rate) was somnolence or sleepiness.

<sup>2-</sup> Plasma cortisol will be obtained prior to leaving the lab for overnight hospital stay and after alcohol cue lab session. Drug plasma concentration will be obtained after alcohol cue lab session.

<sup>3-</sup> Nasal swab for COVID-19 test must be completed 3 days prior to your overnight stay to comply with UCSD-ACTRI's requirement for overnight visits.



Daytime sleepiness may occur that can affect your alertness and motor coordination including impaired driving.

Do not drive, operate heavy machinery, do anything dangerous or do activities that require clear thinking after taking suvorexant. You may still feel drowsy the next day. Do not drive until you feel fully awake.

If you drink alcohol while taking suvorexant, the effects will be increased.

There could be other side effects that we just don't know about yet and we do not know if the same side effects will occur, or if new side effects will emerge in persons who have a problem with alcohol.

The placebo pill will be a pill that looks like real drug but contains no active drug. Study drugs may contain lactose. People who are unable to digest lactose properly are called lactose intolerant. If you are lactose intolerant you might experience side effects such as nausea, abdominal cramping, bloating or gas, after taking study drug. These side effects are usually not dangerous and will stop when the medication is stopped. Please let the study coordinator know if you are lactose intolerant.

#### Alcohol Withdrawal

You must not drink alcohol for at least 2days before the medical clearance at Visit 2. This could put you at risk for alcohol withdrawal symptoms. If you do have alcohol withdrawal symptoms, you will be referred to a local detoxification center. The costs of detoxification will be your responsibility.

## **Alcohol Cue Session Testing Procedures**

Testing procedures could cause unpleasant reactions. You might feel:

- Fatigued (tired) or distressed (anxious or uncomfortable) by the rating scales.
- You will be tempted by your favorite alcoholic beverage and this may give you the urge to drink.
- Depressed or anxious after cue exposure.

### Is there anything else I should know?

- If you are female, you will have a pregnancy test at screening, randomization. Therefore, to participate in the study you must agree to use an effective form of birth control for the study duration.
- If you have been in another research study in the last month, you should tell the study doctor.
- You can't use any drugs or supplements without asking the study doctor.
- We may use information you give us to help find you in case you move. Any information (like your address or phone numbers) will be used only to help find you for follow-up studies.

Blood Sampling: You may feel pain or discomfort when the needle pokes your skin. There may be bruising, swelling, pain, or infection later at the puncture site, although this is unlikely. Dizziness and fainting are possible, but very unlikely. If you have ever felt dizzy or fainted while having blood drawn, you should tell the person drawing your blood. You might not get dizzy if you lie down. If these problems occur, you will be given proper treatment until you recover.

Abnormal Medical Test Results: Medical testing performed during your participation may increase the possibility of receiving an abnormal test result, for example, high blood sugar or elevated liver enzymes.

Version 02/11/2022 



Medical tests performed within the protocol are for research purposes and are not intended to, and may not be suitable for, diagnosing a medical problem. Your medical results will be reviewed by a study physician. Abnormal results will be communicated to you by a research team member. If you decide to pursue medical follow-up, we will release the results to your physician with your written permission. For the Certificate of Confidentiality to protect sensitive information, the identity of the study will not be released to your physician along with the abnormal test results. If you do not have medical insurance, we will supply you with a list of medical service providers in the San Diego area that can be accessed for free or at little cost to you.

Abnormal test results may cause you to experience anxiety and to seek additional medical services, and therefore may be a potential risk of your research participation.

Since alcohol use disorder is an investigational use for suvorexant, there may be some unknown risks that are currently unforeseeable. You will be informed of any significant new findings.

If you choose to join the study, you must agree to take study medication as prescribed and abstain from alcohol for two days in a row before your medical clearance/randomization at Visit #2.

If you are under the influence of alcohol at your appointment, you will have to either stay in our office until your blood alcohol level goes down to .000 on an intoximeter, call someone to pick you up, or call a taxi to take you home at your own expense. If you are found to be impaired by alcohol at your study visit, the visit will have to be rescheduled for another time, and you will not be paid for that visit. Because your blood alcohol level may remain elevated for a period of time after drinking, it is recommended you do not drink for two days before your appointment in order to attain a reading of .000.

# www.ClinicalTrials.gov

Results of this research will not be shared directly with you. A description of this study is available on http://www.ClinicalTrials.gov, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

#### What's in it for me?

You will not benefit personally, but your participation may help identify drugs to help others stop drinking.

### Will I get paid?

Yes, you will be paid \$50 for completing the screening (Visit 1), \$500 for completing randomization/overnight stay/next day laboratorysession (Visit 2), and \$50 for completing the (Visit 3) virtual follow-up. If you complete the study, you will receive a total of \$600. If for any reason you leave the study early, you will be paid only for those study visits that you have completed.

### Will it cost anything to be in the study?

Everything in the study is provided at no cost to you. If you choose to pursue medical follow-up for abnormal medical test results, the financial costs will not be paid by Scripps Research, they will be your responsibility.



## What if I end the study early?

If you quit the study or are taken out early, you will not be paid for follow-up visits you have not completed. You may be asked to return for tests to be sure your health has not changed during the study. The investigator can take you out of the study if you fail to follow study procedures or for other reasons

### What other treatments could I take?

This is not a treatment study. The alternative is not to participate in this study.

# What about confidentiality?

We have several ways to protect electronic data, in both technical ways, as well as by rules and physical security, just as we control access to your paper medical record. Using technology, we hide our computers on the network so that unauthorized viewers can't see them, and these computers can only be accessed with unique passwords and authorization using "security certifications," data encryption in some instances and passwords. We also keep track of who opens what computer files. We give access to members of our research staff on a case-by-case basis for the specific purposes of having them enter data or to help us with your care and our research. We grant this access according to the same level staff would have to look at your medical and research paper files. Thus, we impose a set of standards to protect your information as it resides in our computers.

There also may be other privacy risks that we have not foreseen.

The study doctor, the research staff, and the funding institution will keep your personal information confidential. Your research records could be reviewed by agencies within the Department of Health and Human Services who evaluate and monitor research studies for their accuracy of findings as well as your safety and welfare. These agencies included the Scripps Office for the Protection of Research Subjects (SOPRS), UCSD's Human Research Protections Program, the Food and Drug Administration (FDA) and National Institutes of Health (NIH).

Your privacy will be protected with a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local, civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under the following circumstances: disclosure that a child is being abused, or an indication of intent to hurt yourself or others.

Once this research study is completed, deidentified information or biospecimens collected from you may be stored or used for future research about treatment response.

# What are my rights?

• You can call the staff to ask any questions about this study. The telephone number is listed at the top of this form.



- You can decide not to be in this study, or you can quit after starting. Whatever you do, your medical care at Scripps will not be affected.
- If you have any questions about your rights, call the Scripps Office for the Protection of Research Subjects at (858) 678-6402. You should also read the *Experimental Subject's Bill of Rights*, which is the last page of this form.
- You do not have to be in this study. You still have all your legal rights whether you join the study or not.

### What are my responsibilities if I join?

If you are in this study, you are expected to:

- Follow the instructions of the research staff
- Report any serious or unusual side effects to the study doctor
- Take study drugs as directed
- Keep your study appointments
- Not drink alcohol for 2 days prior to your overnight hospital stay (Visit 2)

## What if I get hurt in the study?

You may call Dr. Shadan at (858) 752-2913, Monday through Friday, 8:00 a.m. to 5:00 p.m., if you get sick or injured while on this study or have any questions about the medication (suvorexant). If you get sick or injured or have questions about the medication at night or on a weekend, you should call Dr. Shadan at (858) 752-2913 or seek treatment at an Urgent Care or Emergency Room facility. If you feel you need immediate attention, you should call 9-1-1.

If you need either medical care or urgent medical treatment as a result of your participation in the study, Scripps Researchgeneral liability insurance will cover these costs.

No money is available to pay you for time off from work. You are not giving up any of your legal rights by being in this study.

### What's in it for the institution and the researchers?

Scripps Research and the study doctor are being paid to do this study by the National Institute on Alcohol Abuse and Alcoholism.

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*

### Suvorexant for Protracted Abstinence in Alcoholism

# I agree to participate.

I have read the explanation of the study and understand it. The study has also been explained to me by Dr. Mason or a member of her research staff. I have had a chance to ask questions and have them answered to my satisfaction. I agree to take part in this study. I have not been forced or made to feel obligated to take part.

I have read the attached Experimental Subject's Bill of Rights, which contains some important information about research studies. I must sign this consent form, the Experimental Subject's Bill of Rights and will be given a signed copy of each to keep.

| Printed Name of Subject | Signature of Subject | | Date |
|---|---|---|---|
| Signature of person conducting the informed consent discussion | | Date | |
| Role of person named above in | the research project | | |



#### \*EXPERIMENTAL SUBJECT'S BILL OF RIGHTS

If I am asked to consent to be a subject in a research study involving a medical experiment, or if I am asked to consent for someone else, I have the right to:

Learn the nature and purpose of the experiment (also called "study" or "clinical trial").

Receive an explanation of the procedures to be followed in the study, and any drug or device to be used.

Receive a description of any discomforts and risks that I could experience from the study.

Receive an explanation of any benefits I might expect from the study.

Learn about the risks and benefits of any other available procedures, drugs or devices that might be helpful to me.

Learn what medical treatment will be made available to me if I should be injured as a result of the study.

Ask any questions about the study or the procedures involved.

Quit the study at any time, and my decision will not be used as an excuse to withhold necessary medical treatment.

Receive a copy of the signed and dated consent form.

Decide to consent or not to consent to a study without feeling forced or obligated.

If I have questions about a research study, I can call the contact person listed on the consent form. If I have concerns about the research staff or need more information about my rights as a subject, I can contact the Scripps Office for the Protection of Research Subjects, which protects volunteers in research studies. I may telephone the Office at (858) 678-6402, 8:00 a.m. to 4:00 p.m. weekdays, or I may write to the Scripps Office for the Protection of Research Subjects c/o Scripps Clinic, Mail Stop SCRC200, 4275 Campus Point Court, Suite 200, San Diego, CA, 92121.

| By signing this document, I agree that I have read ar | nd received a copy of this Bill of Rights. |
|---|---|
| Signature of Subject | Date |
| *California Health & Safety Code, Section 24172 | |

Version 02/11/2022 